CLINICAL TRIAL: NCT06275308
Title: Effect of Raised End-Tidal pCo2 on Choroidal Volume
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Kanwal Nischal, Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY21100163
Record Dates: First submitted 2024-01-24; First posted 2024-02-23 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Intraocular Pressure

STUDY DESIGN:
Intervention Model Description: This is a descriptive case series.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observational Group (Experimental): Manipulation of end tidal carbon dioxide in subjects
  Interventions: Other: Ventilation manipulation

INTERVENTIONS:
Other: Ventilation manipulation — Effects of ventilation manipulation to achieve desired levels of end tidal carbon dioxide

SUMMARY:
This study is to investigate the relationship between arterial carbon dioxide (CO2) concentration and vitreous pressure on the choroidal volume by integrated intraoperative OCT imaging under eye exams under anesthesia.

DETAILED DESCRIPTION:
Children with normal eyes undergoing an exam under anesthesia or a non-intraocular eye procedure will have one eye examined after research consent is taken. Children have very elastic ocular tissues. When they are having an intraocular procedure positive vitreous pressure can cause the iris to prolapse out of the eye and this can cause intraoperative and postoperative complications. The causes of the positive vitreous pressure have been speculated to be due to an increase in choroidal volume. The Choroid is a layer of blood vessels sitting between the sclera and the retina. Ocular Coherence Tomography (OCT) is an imaging tool that allows an optical section of the retina, choroid and sclera to be examined. The subfoveal choroidal thickness has been shown to be a consistent area that can be measured with reliability that the anatomical site of measurement is consistent. By varying the end tidal CO2 the thickness of the choroid will be measured and at the same time the intraocular pressure taken using a pneumatonometer. The OCT is integrated into the operating microscope and is used to take a scan of the fovea. Three scans will be taken after 5minutes of the particular end tidal pCO2. In order to ensure the choroidal thickness is not being influenced by the axial length of the eye, the axial length will be measured using an ultrasound probe at the beginning of the measurements just once. In order to ensure that the position of the head and body is not influencing the choroidal thickness a spirit level will be used to ensure a flat operating bed at the beginning of the measurements.

ELIGIBILITY:
Inclusion Criteria:

* any child undergoing an eye exam under anesthesia for an ophthalmologic reason.
* children between the ages newborn to 8 years of age.

Exclusion Criteria:

* children who are not having an eye exam under anesthesia.
* children with a known medical diagnosis that affect the eye to be studied
* * children over the age of 8 years of age.
* * children with altered cerebral autoregulation, increased intracranial pressure, pulmonary hypertension, or any other condition deemed appropriate by the anesthesiologist.
* children in whom a laryngeal mask airway will not be used

Max Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Intraocular Pressure (IOP) (mmHg) | After induction of anesthesia end tidal CO2 will be manipulated to 40mmHg, then 30mmHg and then 50mmHg. The end tidal CO2 levels will be held for at least 5 minutes after each ventilation manipulation and at the end of this 5 minute period IOP measured
  Measurement of intraocular pressure after maintenance of end tidal pCO2 for 5 minutes at three end tidal pCO2 values : 40mmHg, then 30mmHg and then 50mmHg

SECONDARY OUTCOMES:
Choroidal thickness ( microns) | After induction of anesthesia end tidal CO2 will be manipulated to 40mmHg, then 30mmHg and then 50mmHg. The end tidal CO2 levels will be held for at least 5 minutes after each ventilation manipulation;at the end of 5 minute period choroid images taken
  After 5 minutes of maintenance of end tidal pCO2 at 40mmHg, then 30mmHg and then 50mmHg, ocular coherence tomography (OCT) will be used to capture the subfoveal choroid. The images of the choroid will be provided to blinded individuals who will measure their thickness using the integrated scale on the OCT image.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Monroe, MPH, MBA, Study Director — University of Pittsburgh; Kanwal Nischal, MD,FRCOphth, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No